CLINICAL TRIAL: NCT07012499
Title: The Investigation of Quality of Life and Mental Health Using Remote Monitoring System (Sharesource) With Automated Peritoneal Dialysis in End-stage Renal Disease Patients
Brief Title: QOL and Mental Health Using APD With Remote Monitoring System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-08-0031
Record Dates: First submitted 2025-02-24; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Quality of Life; Mental Health Wellness 1
Keywords: remote control; Automated peritoneal dialysis

STUDY DESIGN:
Intervention Model Description: Comparison of the APD model with internet-based feedback system versus without it
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APD with Sharesource (Experimental): Patients received APD with Sharesource system
  Interventions: Device: Automated peritoneal dialysis with Sharesource device
- APD without Sharesource (Placebo Comparator): Patients received APD without sharesource
  Interventions: Device: APD without sharesource

INTERVENTIONS:
Device: Automated peritoneal dialysis with Sharesource device — Patients receive APD with an FMC device that contains sharesource software which can communicate with the medical team.
  Arms: APD with Sharesource
Device: APD without sharesource — Patients received APD with Same machine but this patients dose not using sharesource software
  Arms: APD without Sharesource

SUMMARY:
Although peritoneal dialysis (PD) is a representative renal replacement therapy along with hemodialysis, number of PD patients decreases every year. Among the various contributing factors for such trends, the essential issue that the patients should perform dialytic therapy by themselves is thought to be critical for the patients to avoid choosing PD as primary dialytic therapy. In particular, unlike hemodialysis, the patients with PD have troubles in getting timely medical advice in their daily life, although continuous advice are essential for maintaining therapy. Thus, remote monitoring and control system is believed to be useful in PD therapy.

Automated PD (APD) is a good option because of its convenience and improved accessibility. So, in Korea, although the rate of incident PD patients was decreased, the proportion of APD were rapidly increased (3.7% in 2001 vs. 39% in 2018, Korean Society of Nephrology (KSN) data) In the COVID-19 pandemic, the investigators should improve Remote therapy monitoring (RTM). Technologies that collect medical information and transmit it to health care providers for patient management, have the potential to improve the patients' outcomes without visiting hospital receiving automated peritoneal dialysis (APD) at home. However, there are only a few retrospective studies and no prospective study about remote patients monitoring programs in APD. Remote medical service is currently illegal in South Korea. However, recently the Korean government has approved remote medical service in only a few areas of Gangwon province, including Wonju city, which belongs to our institution.

Thus, the investigators aim to use such a benefit to investigate the 'Quality of Life (QOL)' in Korean patients undergoing APD. The investigators plan to compare the various clinical indexes, including mainly QOL, mental health focusing depression, and volume-nutritional status between the patients with previous classic APD and APD combined by the SharesourceTM system (Baxter Co.).

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* ESRD patients on APD(≥1 month)
* Consent to participate in the study

Exclusion Criteria:

* Patients who plan to receive kidney transplantation within 1 year
* Patients with co-morbidities: cardiovascular disease(myocardial infarction, heart failure, arrhythmia), cancer, psychiatric diseases, liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of quality of life KDQOL-36 | 6, 12 months
changes of quality of life PHQ-9 | 6, 12 months
changes of quality of life BDI | 6, 12 months
changes of quality of life CESD | 6, 12 months

SECONDARY OUTCOMES:
change volume status | 6, 12 months
  Overhydration (measured by bioimpedance device)
change nutrition status | 6, 12 months
  GNRI (geriatric nutrition risk index), Handgrip strength test (kg)
dialysis adequacy | 6,12 months
  KT/V
Questionnaire form. | 6,12 months
  change of PD perscription, personalized prescription changes, hospital admission, ER admission, unplanned hospital visit, exchanges over telephone
adverse events | 12 months
  peritonitis, mechanical comlications
Body mass index (BMI: kg/m2) | 6 months, 12 months

OTHER OUTCOMES:
Total time or PD | 90 Days
  Total time of PD
Medical coast of treatment | 12 month
  Medical coast

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Kangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No